CLINICAL TRIAL: NCT03589651
Title: A Phase 1b Study of INCMGA00012 in Combination With Other Therapies in Patients With Advanced Solid Tumors
Brief Title: INCMGA00012 in Combination With Other Therapies in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCMGA 0012-102
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Unresectable or Metastatic Solid Tumors
Keywords: Solid tumors; locally advanced unresectable tumor; metastatic solid tumors
MeSH Terms: interventions — epacadostat; parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): INCMGA00012 with epacadostat.
  Interventions: Drug: Retifanlimab; Drug: Epacadostat
- Group B (Experimental): INCMGA00012 with INCB050465.
  Interventions: Drug: Retifanlimab; Drug: INCB050465

INTERVENTIONS:
Drug: Retifanlimab — Part 1: INCMGA00012 at the protocol-defined starting dose administered intravenously every 4 weeks, with dose escalation to determine the maximum tolerated dose.
  Part 2: INCMGA00012 at the recommended dose from Part 1.
Drug: Epacadostat — Part 1: Epacadostat at the protocol-defined starting dose administered orally twice daily, with dose escalation to determine the maximum tolerated dose.
  Part 2: Epacadostat at the recommended dose from Part 1.
  Other Names: INCB024360; INCMGA00012
  Arms: Group A
Drug: INCB050465 — Part 1: INCB050465 at the protocol-defined starting dose administered orally once daily, with dose escalation to determine the maximum tolerated dose. Part 2: INCB050465 at the recommended dose from Part 1.
  Arms: Group B

SUMMARY:
The purpose of this study is to determine the safety, preliminary evidence of clinical activity, and recommended Phase 2 dose (RP2D) of INCMGA00012 in combination with other agents that may improve the therapeutic efficacy of anti-PD-1 monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, locally advanced unresectable or metastatic solid tumors for whom no approved therapy with demonstrated clinical benefit is available or participants who are intolerant to or have declined standard therapy
* Measurable or nonmeasurable tumor lesions per RECIST v 1.1.
* Willing to provide fresh or archival tumor tissue for correlative studies.
* Eastern Cooperative Oncology Group performance status 0 to 1.
* Willingness to avoid pregnancy or fathering children based on protocol-defined criteria.

Exclusion Criteria:

* Receipt of anticancer therapy within 21 days of the first administration of study treatment, with the exception of localized radiotherapy.
* Toxicity of prior therapy that has not recovered to ≤ Grade 1 or baseline (with the exception of alopecia and anemia not requiring transfusional support).
* Laboratory values outside the protocol-defined range at screening.
* Active autoimmune disease requiring systemic immunosuppression in excess of physiologic maintenance doses of corticosteroids.
* Known hypersensitivity to any of the study drugs, excipients, or another monoclonal antibody which cannot be controlled with standard measures (eg, antihistamines and corticosteroids).
* Evidence of interstitial lung disease or active, noninfectious pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | Up to approximately 30 months
  Defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug.

SECONDARY OUTCOMES:
Cmax of INCMGA00012 when given in combination with immune therapies | Up to approximately 4 months
  Defined as maximum observed plasma or serum concentration. Other pharmacokinetic measures (including Cmin and AUC0-t) will also be evaluated.
Tmax of INCMGA00012 when given in combination with immune therapies | Up to approximately 4 months
  Defined as time to maximum concentration. Other pharmacokinetic measures (including Cmin and AUC0-t) will also be evaluated.
Cmax of epacadostat when given in combination with INCMGA00012 | Up to approximately 4 months
  Defined as maximum observed plasma or serum concentration. Other pharmacokinetic measures (including Cmin and AUC0-t) will also be evaluated.
Tmax of epacadostat when given in combination with INCMGA00012 | Up to approximately 4 months
  Defined as time to maximum concentration. Other pharmacokinetic measures (including Cmin and AUC0-t) will also be evaluated.
Cmax of INCB050645 when given in combination with INCMGA00012 | Up to approximately 4 months
  Defined as maximum observed plasma or serum concentration. Other pharmacokinetic measures (including Cmin and AUC0-t) will also be evaluated.
Tmax of INCB050645 when given in combination with INCMGA00012 | Up to approximately 4 months
  Defined as time to maximum concentration. Other pharmacokinetic measures (including Cmin and AUC0-t) will also be evaluated.
Overall response rate | Up to approximately 30 months
  Defined as the percentage of participants having complete response (CR) or partial response (PR) as determined by investigator assessment of radiographic disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and modified RECIST v1.1 for immune-based therapeutics.
Duration of response | Up to approximately 30 months
  Defined as the time from the earliest date of CR or PR until the earliest date at which progression criteria are met or date of death due to any cause, whichever occurs first.
Progression-free survival | Up to approximately 30 months
  Defined as the time from the start of therapy until the earliest date at which progression criteria are met or date of death due to any cause, whichever occurs first.
Overall survival | Up to approximately 30 months
  Defined as the time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Florida - Shands Cancer Center, Gainesville, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Rutgers Cancer Institute of Nj, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Upmc Cancercenter, Pittsburgh, Pennsylvania
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No